CLINICAL TRIAL: NCT06892444
Title: Effects of Sweet Corn Intake on Carotenoid Levels and Gastrointestinal Wellness
Brief Title: Sweet Corn and Carotenoids
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB202500277
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Carotenoids
Keywords: sweet corn; lutein; zeaxanthin; carotenoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yellow Sweet Corn (Experimental): 1.5 cups of yellow sweet corn daily
  Interventions: Dietary Supplement: Yellow Sweet Corn
- White Sweet Corn (Sham Comparator): 1.5 cups of white sweet corn daily
  Interventions: Dietary Supplement: White Sweet Corn

INTERVENTIONS:
Dietary Supplement: Yellow Sweet Corn — Participants will consume 1.5 cups daily of yellow or white canned sweet corn.
  Arms: Yellow Sweet Corn
Dietary Supplement: White Sweet Corn — 1.5 cups daily of canned yellow sweet corn
  Arms: White Sweet Corn

SUMMARY:
This study will assess the effect of daily yellow and white sweet corn intake on serum lutein and zeaxanthin concentrations. Skin carotenoid levels using the Veggie Meter will be assessed, and gastrointestinal symptoms and changes in fecal microbiota during a 4-week intervention period will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Able to provide written consent in English
* Baseline Veggie Meter score of ≤ 250 (Scale from 0 to 850)
* Willing to adhere to study procedures

Exclusion Criteria:

* Baseline Veggie Meter score of >250
* Corn allergy
* Current use of laxatives or antidiarrheal medications
* Previously or currently being treated for intestinal disease, including irritable bowel syndrome, Crohn's disease, ulcerative colitis, celiac disease, or gastrointestinal cancer
* Previous gastrointestinal surgery (e.g., gastric bypass, fundoplication, bowel resection)
* Current cancer treatment
* Current pregnancy
* Vegetarian diet
* Elite athletes or long-distance runners.
* Use of antibiotic drugs within 1 month of the screening visit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of lutein + zeaxanthin | 28 days
  Sum of serum concentrations of lutein and zeaxanthin.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided